CLINICAL TRIAL: NCT07320456
Title: Effect of Longqi Jiangzhi Decoction on Non-alcoholic Fatty Liver Disease: a Randomized Clinical Trial
Brief Title: A Clinical Trial of Longqi Jiangzhi Decoction Against Non-alcoholic Fatty Liver Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LJD2025001
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The control placebo is a ten-fold dilution of the Longqi Jiangzhi decoction, supplemented with colorants and bittering agents to mimic the appearance and color of the treatment drug. An independent researcher (not involved in the trial operations or evaluations) is responsible for managing the randomization sequence and drug coding, and will distribute the appropriate drugs to participants at the right times. This ensures that the trial operators and evaluators are unaware of the treatment type; only the independent researcher has this knowledge. During the experiment, the assessment of treatment effects and the recording of adverse events are carried out by independent evaluators who are unaware of the treatment groups. Both the trial operators and the evaluators do not have access to the drug coding and randomization sequence.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): These medicines of Longqi Jiangzhi decoction are uniformly decocted, prepared, and packaged by the Pharmacy of Shanghai Municipal Hospital of Traditional Chinese Medicine. The administration is oral, taken twice daily, one packet each time, for a treatment period of 8 weeks. In addition, following the guidelines, all participants will receive lifestyle interventions, including diet and exercise health education before enrollment to ensure calorie control and exercise compliance.
  Interventions: Drug: Longqi Jiangzhi decoction
- Control group (Placebo Comparator): These placebo medicines are uniformly decocted, prepared, and packaged by the Pharmacy of Shanghai Municipal Hospital of Traditional Chinese Medicine. The administration is oral, taken twice daily, one packet each time, for a treatment period of 8 weeks. In addition, following the guidelines, all participants will receive lifestyle interventions, including diet and exercise health education before enrollment to ensure calorie control and exercise compliance.
  Interventions: Drug: Control placebo

INTERVENTIONS:
Drug: Longqi Jiangzhi decoction — Below is the composition of Longqi Jiangzhi decoction: Gentiana Scabra 5g, Astragalus membranaceus 10g, Rhizoma Alismatis 10g, Crataegus pinnatifida 10g, Citri Reticulatae Pericarpium 5g.
  Arms: Treatment group
Drug: Control placebo — The control placebo is a ten-fold dilution of the Longqi Jiangzhi decoction, supplemented with colorants and bittering agents to mimic the appearance and color of the treatment drug.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if Longqi Jiangzhi decoction works to treat non-alcoholic fatty liver disease in adults. It will also learn about the safety of drug Longqi Jiangzhi decoction. Researchers will compare drug Longqi Jiangzhi decoction to a placebo (a look-alike substance that contains no drug) to see if drug Longqi Jiangzhi decoction works to treat non-alcoholic fatty liver disease. Participants will: Take drug Longqi Jiangzhi decoction or a placebo every day for eight weeks Keep a record of their symptoms and the degree of hepatic steatosis before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years, both genders eligible;
2. Meets the diagnostic criteria for NAFLD;
3. Meets the diagnostic criteria for Traditional Chinese Medicine Spleen Deficiency and Damp-Heat Syndrome;
4. Has significant risk factors: CAP≥238dB/m, Body Mass Index (BMI) ≥23 kg/m²;
5. Has not received any anti-NAFLD medication treatment in the past month;
6. Normal major organ function, including heart, kidney, and liver functions, specifically: no significant abnormalities on electrocardiogram; normal serum creatinine and urea nitrogen; normal serum bilirubin and albumin levels;
7. Has sufficient cognitive and understanding abilities to comprehend the study content and its potential risks and benefits;
8. Voluntarily participates in the study and signs an informed consent form.

Exclusion Criteria:

1. Has liver steatosis due to other definitive causes, such as alcoholic liver disease, drug-induced liver injury, viral hepatitis infections (e.g., hepatitis B, hepatitis C, etc.);
2. Has other serious liver diseases, such as autoimmune liver diseases, primary biliary cholangitis, Wilson's disease, etc.;
3. Has severe dysfunction of major organs such as the heart, kidneys, lungs, etc., such as severe heart failure (NYHA functional classification III or above), renal failure (glomerular filtration rate eGFR < 30 mL/min/1.73m²), acute exacerbation of chronic obstructive pulmonary disease, etc.;
4. Has other serious systemic diseases, such as malignant tumors, active systemic lupus erythematosus, etc.;
5. Known allergy or intolerance to any component of the study medication;
6. Has participated in another clinical trial within the last three months;
7. Pregnant women, lactating women, or women of childbearing age who refuse to use effective contraception during the trial;
8. Has severe mental illness or behavioral disorders that may affect adherence to the study protocol;
9. Other conditions that the researcher considers unsuitable for participation in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
controlled attenuation parameter | through study completion, an average of 8 weeks
  A liver fiber diagnostic instrument (Fibro Touch) is used to perform instantaneous elastic hardness testing. The controlled attenuation parameter usually represents liver fat content, whereas higher scores mean a worse outcome.

SECONDARY OUTCOMES:
body weight | through study completion, an average of 8 weeks
  weighing on a scale
total cholesterol | through study completion, an average of 8 weeks
  serum biochemistry
triglyceride | through study completion, an average of 8 weeks
  serum biochemistry
fasting plasma glucose | through study completion, an average of 8 weeks
  serum biochemistry
alanine aminotransferase | through study completion, an average of 8 weeks
  serum biochemistry
aspartate aminotransferase | through study completion, an average of 8 weeks
  serum biochemistry

OTHER OUTCOMES:
urea nitrogen | through study completion, an average of 8 weeks
  serum biochemistry
creatinine | through study completion, an average of 8 weeks
  serum biochemistry

IPD SHARING:
Plan to Share IPD: Undecided